CLINICAL TRIAL: NCT00581490
Title: Biochemical and Radiological Indicators of Cardiovascular Morbidity in Children With Premature Pubarche
Acronym: PP
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 030292
Record Dates: First submitted 2007-12-20; First posted 2007-12-27 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Evidence of Cardiovascular Morbidity
Keywords: Premature pubarche; Adrenal hyperandrogenism; Metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA sample from consented subjects and controls
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Idiopathic premature pubarche: Children with premature pubarche without precious puberty, adrenal hyperplasia or androgen secreting tumors

SUMMARY:
Children with premature pubarche will have radiological and radial artery tonometry evidence of cardiovascular morbidity at diagnosis when compared to matched controls.

DETAILED DESCRIPTION:
Premature pubarche (PP), also called premature adrenarche (PA), is the early appearance of pubic hair before the age of 8 in girls and before 9 in boys. It had been shown that PP results from excess adrenal androgens. The terms PP and PA are used synonymously and differ from premature (precocious) puberty, the early activation of hypothalamic-pituitary gonadal axis. The incidence of PP is almost tenfold higher in girls than in boys. PP in the absence of congenital adrenal hyperplasia, virilizing ovarian or adrenal tumors has been regarded in the past as a benign phenomenon that may be associated with transient acceleration of growth and bone maturation and was not thought to have an adverse effect on the onset and progression of puberty and on final height in most patients. However, recent evidence suggests that hyperinsulinemia and obesity are common features in prepubertal and pubertal girls with a history of PP. Peri- and post-pubertal girls with PP exhibit an increase in incidence of hirsutism and polycystic ovary syndrome (PCOS). PCOS, a common hyperandrogenic disorder of women, is characterized by functional ovarian hyperandrogenism (FOH). FOH is defined as a 17-hydroxyprogesterone and/or androstenedione level >2 SD above that of the mean for control subjects after subcutaneous gonadotropin-releasing hormone agonist (GnRHa) stimulation during dexamethasone suppression of the adrenal glands. An increased risk of ovulatory dysfunction and FOH in adolescence detectable 3 years after menarche has also been reported in children diagnosed with PP. Serum triglyceride levels in premature adrenarche patients are higher when compared to controls throughout all stages of pubertal development. Boys with PP show reduced insulin sensitivity, independent of obesity, as observed in girls with PP. In Hispanic and Caribbean girls studies have shown prenatal influence on the development of PP. The lowest birth weights are found in this group of girls with PP who also have pronounced hyperinsulinism. Also, the presence of dyslipidemia in girls with PP depends on weight gain after birth. It has been shown that prepubertal girls are inherently more insulin resistant than boys which has been suggested to be related to the intrinsic difference in sex linked genes. Early metformin therapy prevents progression from PP to PCOS in a high risk group of former low birth weight girls, supporting the key role of insulin resistance in the ontogeny of PCOS.

Early intervention in PP can be initiated before marked obesity, diabetes, hypertension and increased cardiovascular morbidity related to insulin resistance become associated with endothelial dysfunction and abnormal vascular structure. Any intervention to decrease cardiovascular morbidity and mortality related to obesity and insulin resistance optimally begins in childhood. The short term goal of this proposal is to collect non-invasive evidence of cardiovascular disease morbidity risk factors at the time of PP diagnosis and to determine how they progress. Symptomatic endpoints used in most adult intervention trials, i.e. cardiac events and death, are not applicable in the setting of childhood disease.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls with isolated premature pubarche

Exclusion Criteria:

* Congenital adrenal hyperplasia
* Precocious puberty
* Androgen producing tumors

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Boys below the age of 9; girls below the age of 8 if Caucasian and below age 6 if African American
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2003-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Changes in biometric and radiological features between subjects and matched controls | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Revi P. Mathew, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States